CLINICAL TRIAL: NCT04555226
Title: Randomized Controlled Trial of the Efficacy of Lymph Node Dissection on Stage IIICr of Cervical Cancer
Brief Title: The Efficacy of Lymph Node Dissection for Stage IIICr of Cervical Cancer(CQGOG0103)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Jiangxi Provincial Cancer Hospital (Other); Anhui Provincial Cancer Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Hebei Medical University Fourth Hospital (Other); Zhejiang Cancer Hospital (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Qilu Hospital of Shandong University (Other); Fujian Cancer Hospital (Other Government); Sichuan Cancer Hospital and Research Institute (Other); Cancer Hospital of Guizhou Province (Other); West China Second University Hospital (Other); Tongji Hospital (Other); The Affiliated Ganzhou Hospital of Nanchang University (Other); First Affiliated Hospital of Gannan Medical University (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); Third Affiliated Hospital of Xinjiang Medical University (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Fujian Maternity and Child Health Hospital (Other); Shandong Cancer Hospital and Institute (Other); Sun Yat-sen University Cancer Hosptial (Unknown)
Responsible Party: Principal Investigator, Dongling Zou, Director of Gynecologic Oncology Department, Chongqing University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG0103
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cervical Cancer
Keywords: Stage IIICr of cervical cancer; Lymph node dissection; Chemoradiation; PFS
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment group (Active Comparator): Standard chemoradiation (Pelvic EBRT/Extended-field EBRT + concurrent platinum-containing chemotherapy + brachytherapy±pembrolizumab).
  Interventions: Radiation: Standard chemoradiation±pembrolizumab
- Experimental group (Experimental): Open/minimally invasive pelvic and para-aortic lymph node dissection followed by chemoradiation (Pelvic EBRT/Extended-field EBRT + concurrent platinum-containing chemotherapy + brachytherapy±pembrolizumab).
  Interventions: Procedure: Lymph node dissection; Radiation: Chemoradiation± pembrolizumab

INTERVENTIONS:
Procedure: Lymph node dissection — Open/minimaly invasive pelvic and para-aortic lymph node dissection
  Arms: Experimental group
Radiation: Standard chemoradiation±pembrolizumab — 1. A point/HCR-CTV D90≥80Gy(+20%).2. Extended-field EBRT: image-positive common iliac LN with SD≥10mm and/or image-positive PALN.3. Target doses for the image-positive nodes can range from 55 to 60Gy.4. Concurrent 5 cycles platinum-containing chemotherapy(Cisplatin 40mg/m2 q1w or Carboplatin AUC=2 q1w).5. CCRT will be completed in 56 days.6. The patients who received combined immunotherapy were treated with pembrolizumab (200mg, q3w, 3 cycles) during CCRT.7.After CCRT if the cervix biopsy shows residual tumor and/or imaging indicates that there are still positive LN with SD≥15mm in the pelvic and abdominal cavity, 3 cycles adjuvant chemotherapy (TAX 135mg/m2, DDP 50mg/m2, q3w or TAX 135mg/m2, CBP AUC=4, q3W) ± brachytherapy (if point A or HR-CTV D90 < 96Gy) ± pembrolizumab(suitable for the patients who combined immunotherapy,200mg, q3w, 3 cycles) will be performed.8.Maintenance treatment with pembrolizumab (400mg, q6w) is optional for the combined immunotherapy patiants.
  Arms: Standard treatment group
Radiation: Chemoradiation± pembrolizumab — 1. A point/HCR-CTV D90≥80Gy(+20%).2. Extended-field EBRT: image-positive common iliac LN with SD≥10mm and/or image-positive PALN.3. Target doses for the image-positive nodes can range from 55 to 60Gy.4. Concurrent 5 cycles platinum-containing chemotherapy(Cisplatin 40mg/m2 q1w or Carboplatin AUC=2 q1w).5. CCRT will be completed in 56 days.6. The patients who received combined immunotherapy were treated with pembrolizumab (200mg, q3w, 3 cycles) during CCRT.7.After CCRT if the cervix biopsy shows residual tumor and/or imaging indicates that there are still positive LN with SD≥15mm in the pelvic and abdominal cavity, 3 cycles adjuvant chemotherapy (TAX 135mg/m2, DDP 50mg/m2, q3w or TAX 135mg/m2, CBP AUC=4, q3W) ± brachytherapy (if point A or HR-CTV D90 < 96Gy) ± pembrolizumab(suitable for the patients who combined immunotherapy,200mg, q3w, 3 cycles) will be performed.8.Maintenance treatment with pembrolizumab (400mg, q6w) is optional for the combined immunotherapy patiants.
  Arms: Experimental group

SUMMARY:
This is an national, prospective, multicenter and randomized clinical study designed to determine if patients with stage IIICr of cervical cancer have longer PFS and/or OS with lymph node dissection before CCRT when compared to CCRT.

DETAILED DESCRIPTION:
All eligible patients will be equally randomized between the 2 following treatment groups (stratified factors: whether para-aortic lymph nodes were image-positive):

Standard treatment group: standard chemoradiation (Pelvic EBRT/Extended-field EBRT + concurrent platinum-containing chemotherapy+brachytherapy ±pembrolizumab).

Experimental group: open/minimally invasive pelvic and para-aortic lymph node dissection followed by chemoradiation±pembrolizumab. (Level of lymph node dissection: At least the inferior mesenteric artery. Chemoradiation ±pembrolizumab will be performed postoperatively within 28 days.)

ELIGIBILITY:
Inclusion Criteria:

1. Histopathology: squamous cell carcinoma, adenocarcinoma, adeno-squamous cell carcinoma
2. Cervical cancer stage IIICr (confirmed by CT/MRI/PET/CT) and the short diameter of image-positive lymph node ≥15mm
3. ECOG score 0~1
4. Expected survival over 6 months
5. The serum or urine pregnancy test must be negative within 7 days before enrollment for the women of childbearing age who should agree that contraception must be used during the trial
6. No surgical contraindication

Exclusion Criteria:

1. Activity or uncontrol severe infection
2. Active hepatitis B, Liver cirrhosis, Decompensated liver disease
3. History of immune deficiency, including HIV positive or suffering from other immunodeficiency disease
4. Active autoimmune disease requiring systemic treatment (e.g., use of disease-modifying medications, corticosteroids, or immunosuppressive medications). Replacement therapies (e.g., thyroxine, insulin, or physiological corticosteroid replacement for adrenal or pituitary insufficiency) were not counted as systemic therapies, and subjects were permitted to use these therapies
5. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
6. Chronic renal insufficiency or renal failure
7. Has combined with other malignant tumor which diagnosed within 5 years and/or needed to be treated
8. Myocardial infarction, severe arrhythmia and NYHA (New York heart association)≥2 for congestive heart failure
9. Has had an allogenic tissue/solid organ transplant
10. A history of pelvic artery embolization
11. A history of pelvic radiotherapy
12. A history of partial hysterectomy or radical hysterectomy
13. A history of immunotherapy or undergoing immunotherapy
14. A history of severe allergic reactions to platinum-based chemotherapy drugs, pembrolizumab and/or any excipients
15. During the treatment for complications, the drugs which lead to serious liver and/or kidney function impairment need to be used, such as tuberculosis

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  Progression-free survival

SECONDARY OUTCOMES:
OS | 3 and 5 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Dongling Zou, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Sanjose S, Serrano B, Castellsague X, Brotons M, Munoz J, Bruni L, Bosch FX. Human papillomavirus (HPV) and related cancers in the Global Alliance for Vaccines and Immunization (GAVI) countries. A WHO/ICO HPV Information Centre Report. Vaccine. 2012 Nov 20;30 Suppl 4:D1-83, vi. doi: 10.1016/S0264-410X(12)01435-1. No abstract available. PMID 23510764
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Jolly S, Uppal S, Bhatla N, Johnston C, Maturen K. Improving Global Outcomes in Cervical Cancer: The Time Has Come for International Federation of Gynecology and Obstetrics Staging to Formally Incorporate Advanced Imaging. J Glob Oncol. 2018 Sep;4:1-6. doi: 10.1200/JGO.2016.007534. Epub 2017 Mar 21. No abstract available. PMID 30241155
- [Background] Bhatla N, Berek JS, Cuello Fredes M, Denny LA, Grenman S, Karunaratne K, Kehoe ST, Konishi I, Olawaiye AB, Prat J, Sankaranarayanan R, Brierley J, Mutch D, Querleu D, Cibula D, Quinn M, Botha H, Sigurd L, Rice L, Ryu HS, Ngan H, Maenpaa J, Andrijono A, Purwoto G, Maheshwari A, Bafna UD, Plante M, Natarajan J. Revised FIGO staging for carcinoma of the cervix uteri. Int J Gynaecol Obstet. 2019 Apr;145(1):129-135. doi: 10.1002/ijgo.12749. Epub 2019 Jan 17. PMID 30656645
- [Background] Goff BA, Muntz HG, Paley PJ, Tamimi HK, Koh WJ, Greer BE. Impact of surgical staging in women with locally advanced cervical cancer. Gynecol Oncol. 1999 Sep;74(3):436-42. doi: 10.1006/gyno.1999.5472. PMID 10479506
- [Background] Kohler C, Mustea A, Marnitz S, Schneider A, Chiantera V, Ulrich U, Scharf JP, Martus P, Vieira MA, Tsunoda A. Perioperative morbidity and rate of upstaging after laparoscopic staging for patients with locally advanced cervical cancer: results of a prospective randomized trial. Am J Obstet Gynecol. 2015 Oct;213(4):503.e1-7. doi: 10.1016/j.ajog.2015.05.026. Epub 2015 May 15. PMID 25986030
- [Background] Gouy S, Morice P, Narducci F, Uzan C, Martinez A, Rey A, Bentivegna E, Pautier P, Deandreis D, Querleu D, Haie-Meder C, Leblanc E. Prospective multicenter study evaluating the survival of patients with locally advanced cervical cancer undergoing laparoscopic para-aortic lymphadenectomy before chemoradiotherapy in the era of positron emission tomography imaging. J Clin Oncol. 2013 Aug 20;31(24):3026-33. doi: 10.1200/JCO.2012.47.3520. Epub 2013 Jul 15. PMID 23857967
- [Background] Dag Z, Yilmaz B, Dogan AK, Aksan DU, Ozkurt H, Kizilkaya HO, Arslan D. Comparison of the prognostic value of F-18 FDG PET/CT metabolic parameters of primary tumors and MRI findings in patients with locally advanced cervical cancer treated with concurrent chemoradiotherapy. Brachytherapy. 2019 Mar-Apr;18(2):154-162. doi: 10.1016/j.brachy.2018.11.005. Epub 2018 Dec 26. PMID 30594422
- [Background] Frumovitz M, Querleu D, Gil-Moreno A, Morice P, Jhingran A, Munsell MF, Macapinlac HA, Leblanc E, Martinez A, Ramirez PT. Lymphadenectomy in locally advanced cervical cancer study (LiLACS): Phase III clinical trial comparing surgical with radiologic staging in patients with stages IB2-IVA cervical cancer. J Minim Invasive Gynecol. 2014 Jan-Feb;21(1):3-8. doi: 10.1016/j.jmig.2013.07.007. Epub 2013 Jul 31. PMID 23911560
- [Background] Gold MA, Tian C, Whitney CW, Rose PG, Lanciano R. Surgical versus radiographic determination of para-aortic lymph node metastases before chemoradiation for locally advanced cervical carcinoma: a Gynecologic Oncology Group Study. Cancer. 2008 May 1;112(9):1954-63. doi: 10.1002/cncr.23400. PMID 18338811
- [Background] Cho WK, Kim YI, Park W, Yang K, Kim H, Cha H. Para-aortic lymph node recurrence after curative radiotherapy for cervical cancer. Int J Gynecol Cancer. 2019 Sep;29(7):1116-1120. doi: 10.1136/ijgc-2019-000615. PMID 31474588
- [Background] Cosin JA, Fowler JM, Chen MD, Paley PJ, Carson LF, Twiggs LB. Pretreatment surgical staging of patients with cervical carcinoma: the case for lymph node debulking. Cancer. 1998 Jun 1;82(11):2241-8. doi: 10.1002/(sici)1097-0142(19980601)82:113.0.co;2-t. PMID 9610705
- [Derived] He M, Guo M, Zhou Q, Tang Y, Zhong L, Liu Q, Fan X, Zhao X, Zhang X, Chen G, Shen Y, Xu Q, Chen X, Li Y, Zou D. Efficacy of lymph node dissection on stage IIICr of cervical cancer before CCRT: study protocol for a phase III, randomized controlled clinical trial (CQGOG0103). J Gynecol Oncol. 2023 May;34(3):e55. doi: 10.3802/jgo.2023.34.e55. Epub 2023 Mar 23. PMID 36998225